CLINICAL TRIAL: NCT06875999
Title: The Effect of Pet Therapy on Pain, Emotional Symptoms and Physiological Parameters in Children Who Underwent Allergy Testing; Randomized Controlled Study
Brief Title: Pet Therapy Effects on Pain, Emotional and Physiological Responses in Children Undergoing Allergy Testing
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mehtap METİN KARAASLAN (Other)
Responsible Party: Sponsor-Investigator, Mehtap METİN KARAASLAN, ASSIST. PROF., Recep Tayyip Erdogan University
Organization: Recep Tayyip Erdogan University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Allergy skin test
Record Dates: First submitted 2025-03-12; First posted 2025-03-14 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Allergy Testing; Pain, Emotional Symptoms and Physiological Parameters
Keywords: Allergy Testing; Children; Animal-Assisted Therapy; Emotions
MeSH Terms: conditions — Pain | interventions — Animal Assisted Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: Routine clinical practice (No Intervention): In the control group, the Personal Information Form, FLACC Pain Scale and Children's Emotional Indicator Scale (CEMS) will be completed and physiologic parameters will be recorded (pre-procedure). Routine tests will be performed by equipped nurses on the inner side of the forearm, 5 cm from the wrist and 3 cm from the antecubital fossa, in the skin area with intact skin integrity. After the procedure, CEMS and FLACC Pain Scale will be filled again and physiologic parameters will be recorded.
- Animal-assisted therapy: fish in a fishbowl and the red fish song (Experimental): In the intervention group, the Personal Information Form, FLACC pain scale, and Children's Emotional Indicator Scale (CEMS) will be completed and physiologic parameters will be recorded (pre-procedure). Children will be allowed to communicate with fish before the procedure starts. During the procedure, the tests will be performed by equipped nurses on the inner side of the forearm, 5 cm from the wrist and 3 cm from the antecubital fossa, in the skin area with intact skin integrity, with the betta fish still next to it. After the procedure, CEMS and FLACC pain scale will be filled again and physiologic parameters will be recorded.
  Interventions: Behavioral: animal assisted therapy

INTERVENTIONS:
Behavioral: animal assisted therapy — The Children's Emotional Indicator Scale (Facial expression, Vocalization, Activity, Interaction and Cooperation Level) will be used to provide a simple, objective and consistent method to determine children's emotional behavior during stressful medical procedures. The FLACC scale will be used for pain. In addition, all physiological parameters including pulse rate, saturation value and respiration will be measured and recorded with a pulse oximeter device. Animal assisted therapy will be applied to the participants in the study group to reduce the stress of the children. In animal-assisted therapy, the child will be shown a fish in a glass bowl and a red fish song will accompany the process. In the study, participant children will be randomly assigned to intervention and control groups.
  Arms: Animal-assisted therapy: fish in a fishbowl and the red fish song

SUMMARY:
In recent decades, the prevalence of allergic diseases, particularly respiratory allergies, has risen significantly. In childhood, house dust mites are the primary indoor allergen in infancy, while the prevalence of pollen sensitization increases with age. As one of the largest immunologic organs, the skin frequently displays allergic responses; therefore, the Skin Prick Test (SPT) is widely used for diagnostic purposes. SPT is quick, cost-effective, highly sensitive, and rarely causes adverse effects, yet it may still induce stress or anxiety in children-especially younger ones or when applied on the back.

Although distraction methods (e.g., toys, games, DistrACTION® Cards) are commonly used to reduce discomfort in minimally invasive pediatric procedures, there is limited research on strategies to alleviate stress during SPT. This randomized controlled trial (RCT) aims to investigate the impact of pet therapy using betta fish on children's emotional symptoms (such as anger or irritability) and physiological parameters during SPT. The study will include 80 children, aged 3-6, who attend a pediatric allergy clinic between April 2025 and April 2026. Participants will be randomly assigned to control or experimental groups through simple and block randomization, ensuring age balance. Data collection instruments include a Personal Information Form, the Children's Emotional Indicator Scale, FLACC Pain Scale, and a Physiological Parameter Monitoring Form.

The study posits two main hypotheses:

Pet therapy positively affects emotional indicators of children based on their age.

Pet therapy influences physiological parameters by age group. Findings from this research may inform evidence-based interventions to reduce stress and anxiety in pediatric patients undergoing minimally invasive procedures like SPT.

DETAILED DESCRIPTION:
In recent years, there has been a marked increase in the prevalence of allergic diseases. In particular, the incidence of allergic respiratory diseases has almost doubled in the last two decades. This increase is thought to be related to increased sensitization to both indoor and outdoor allergens. Indoors, house dust mites remain the most important cause of allergic sensitization in infants. With increasing age, the prevalence of aeroallergens, especially pollen, increases and sensitization to indoor and outdoor allergens reaches similar levels around three years of age. Sensitization to both allergen groups also increases during childhood. In addition to aeroallergens, there is also immune sensitization to foodborne and drug allergens. The skin is one of the largest immunologic organs, the most frequent target of allergic responses and responds to a wide range of allergic agents. Skin prick test (SPT) is a sensitive method to investigate these allergic disorders. When antigen combines with immunoglobulin E (IgE) antibodies fixed to mast cells, chemical mediators are released from mast cells within five minutes, resulting in the formation of a wheal. SPT is a rapid, simple, low-cost, easy-to-apply and highly sensitive diagnostic method to assess environmental allergy sensitization. This method has high sensitivity and positive predictive ability. Compared with the specific IgE blood test, the accuracy of the test is over 95% and side effects are very rare. SPT can generally be performed without discomfort and a large proportion of patients can tolerate this test without distress. However, the nature of the procedure may cause stress and anxiety, especially in children. Minimally invasive procedures such as venipuncture, dental treatment and routine vaccinations may cause discomfort in children and distraction methods are used in these cases. There is limited information on the effects of SPT on pain and anxiety in children. Existing studies have generally focused on fear and anxiety. Karaatmaca et al. (2021) found that mothers had higher pre-test and post-test STAI anxiety scores than fathers and that parental gender had a significant effect on anxiety. In addition, SPT was found to cause anxiety and pain in some children, especially at young ages and when applied on the back. In a study by Erdim (2022), the use of DistrACTION® Cards to distract children aged 6-10 years during a skin puncture test was examined. In this study, it was found that the pain scores of children during and after the procedure were significantly lower compared to the control group and the use of DistrACTION Cards was effective in reducing the pain and anxiety levels of children. Since the emotional indicators of children have never been evaluated during allergy testing, which is a minimally invasive procedure, this study was planned as a randomized controlled trial to determine the effect of pet therapy application on emotional symptoms and physiological parameters according to age periods in children during allergy testing.

Hypotheses of the study; H1a: Pet therapy has an effect on pain and emotional indicators of children according to their age periods.

H1b: Pet therapy has an effect on the physiological parameters of the child according to age periods.

This study was planned as a randomized controlled trial to determine the effect of pet therapy application on emotional symptoms and physiological parameters according to age periods in children during allergy testing. It included children between the ages of 3-6 who applied to the pediatric allergy outpatient clinics of a training and research hospital between April 2025 and April 2026 and underwent allergy testing. The research sample will consist of children who applied to the pediatric allergy outpatient clinics on the specified dates, met the research criteria and volunteered to participate in the study. Dependent t test analysis was taken into consideration in sample size calculation. With a Type I error rate of 5%, effect size (ES) and moderate power (ES=0.25) of 99%, it was calculated that a total of at least 80 children, 40 children in each group, should be included in the study. In the study, "simple randomization and block randomization methods" will be used to assign participants to control and experimental groups. Numbers will be assigned to the experimental and control groups on www.randomizer.org and blocking will be done according to age to ensure balance between the groups. Personal Information Form, Children's Emotional Indicator Scale, FLACC Pain Scale and Physiological Parameter Monitoring Form will be used to collect the data. Betta fish will be used as the intervention tool in the study.

ELIGIBILITY:
Inclusion Criteria:

* No previous allergy testing
* 3-6 years old
* Stable hemodynamics
* No chronic disease
* The child has no intellectual or neurological disability
* The mother has no obstacle to communication
* Mother is literate
* Families and children agree to participate in the study.

Exclusion Criteria:

* The child does not meet the inclusion criteria
* The mother does not meet the inclusion criteria
* Child's and mother's unwillingness to participate in the study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
reduce children's stress and pain during allergy testing | one year
  Children's pain and stress during the procedure were measured using validated scales or physiological parameters. CEMS consists of five categories of observable emotional behaviors (Facial expression, Vocalization, Activity, Interaction, and Level of cooperation). Each category has a value between 1-5. The total score that can be obtained from the scale varies between 5-25. The higher the scores obtained from the scale, the higher the negative emotional indicators. FLACC Pain Scale is used in awake patients by observation for 1 to 5 minutes. The scale consists of five elements: face, leg, movement, crying, activity status and degree of consolability. Each category is evaluated between 0-2, the total score ranges from 0 to 10. A score of 0 indicates that the child is calm and relaxed, a score of 1-3 indicates that the child is mildly uncomfortable, scores between 4-6 indicate that the child has moderate pain, and a score of 7-10 indicates severe pain.

IPD SHARING:
Plan to Share IPD: Undecided
The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

REFERENCES:
- [Background] Yazici S, Gunes S, Kurtulus-Cokboz M, Kemer O, Baranli G, Asik-Akman S, Can D. Allergen variability and house dust mite sensitivity in pre-school children with allergic complaints. Turk J Pediatr. 2018;60(1):41-49. doi: 10.24953/turkjped.2018.01.006. PMID 30102478
- [Background] Bains P, Dogra A. Skin prick test in patients with chronic allergic skin disorders. Indian J Dermatol. 2015 Mar-Apr;60(2):159-64. doi: 10.4103/0019-5154.152513. PMID 25814704
- [Background] Erdim L. The effect on pain and anxiety levels of using DistrACTION(R) Cards to distract children during a skin-prick test: a randomized controlled experimental study. Minerva Pediatr (Torino). 2022 Apr;74(2):167-175. doi: 10.23736/S2724-5276.21.06008-0. Epub 2021 Apr 2. PMID 33820412
- [Background] Karaatmaca B, Sahiner UM, Soyer O, Sekerel BE. The impact of skin prick testing on pain perception and anxiety in children and parents. Allergol Immunopathol (Madr). 2021 Mar 1;49(2):72-79. doi: 10.15586/aei.v49i2.68. eCollection 2021. PMID 33641297